CLINICAL TRIAL: NCT06810505
Title: A Phase 3, Multicenter, 12-Week, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Atogepant for the Preventive Treatment of Chronic Migraine in Pediatric Subjects 12 to 17 Years of Age
Brief Title: A Study of Oral Atogepant Tablets to Assess Adverse Events and Change in Disease Activity To Prevent Migraine in Participants Aged 12 to 17 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-712; 2024-513836-28
Record Dates: First submitted 2025-01-31; First posted 2025-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Migraine
Keywords: Migraine; Chronic Migraine; Atogepant; QULIPTA; AQUIPTA
MeSH Terms: conditions — Migraine Disorders | interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atogepant (Experimental): Participants will receive atogepant once daily for 12 weeks.
  Interventions: Drug: Atogepant
- Placebo for Atogepant (Placebo Comparator): Participants will receive placebo for atogepant once daily for 12 weeks.
  Interventions: Drug: Placebo for Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral tablet
  Other Names: Qulipta; Aquipta
  Arms: Atogepant
Drug: Placebo for Atogepant — Oral tablet
  Arms: Placebo for Atogepant

SUMMARY:
Migraine is a disease that most often causes moderate to severe headache on one side of the head. A migraine attack is a headache that may be accompanied by throbbing, nausea, vomiting, sensitivity to light and sound, or other symptoms. The goals of the study are to evaluate adverse events and how well treatment of atogepant works compared to placebo (looks like the study treatment but contains no medicine) in preventing chronic migraine in participants between 12 and 17 years of age.

Atogepant is a medicine currently approved in the United States and Europe for the preventive treatment of migraine in adult patients with migraine and is being studied for the preventative treatment of chronic migraine in participants between the ages of 12 and 17 years. Participants will be randomly assigned to one of the 2 groups to be treated with either atogepant or placebo. This study is double-blinded, which means that neither the patients nor the study doctors know who is given which study treatment. Approximately 420 participants 12 to 17 years of age with chronic migraine will be enrolled at approximately 70 sites across the world.

Participants will receive oral tablets of atogepant or placebo once daily for 12 weeks and will be followed for 4 weeks.

Participants will attend regular visits during the study at a hospital or clinic and the effects of treatment will be checked by completion of a daily diary, medical assessments, blood tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3) (2018) for at least 6 months as of Visit 1.
* During the last 28 days of the screening/baseline period, and as per eDiary:

  * Participant must have completed the eDiary for a minimum of 20 out of 28 days.
  * Participant has >= 15 headache days.
  * Participant has >= 8 migraine days.

Exclusion Criteria:

* Clinically significant hypertension per investigator's judgment.
* History of any clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, cardiovascular or neurologic disease.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 16 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Change From Baseline in Mean Monthly Migraine Days | Baseline (Week 0) through Week 12
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.

SECONDARY OUTCOMES:
Change From Baseline in Mean Monthly Headache Days | Baseline (Week 0) through Week 12
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication (e.g., ibuprofen, triptan) was used after the start of the headache, in which case no minimum duration will be specified. Calendar days begin at midnight and last until 11:59 PM.
Change From Baseline in Mean Monthly Acute Medication Use Days | Baseline (Week 0) through Week 12
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
Percentage of Participants who Achieve at Least a 50% Reduction in 3-month Average of Monthly Migraine Days | Baseline (Week 0) through Week 12
  A migraine day is defined as any calendar day on which a migraine occurs as per participant eDiary. Calendar days begin at midnight and last until 11:59 PM.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL) Total Score | Baseline (Week 0) through Week 12
  The PedsQL is a 23-item measure that evaluates quality of life in four areas of functioning: physical, emotional, social, and school functioning. The PedsQL yields a total quality of life score and two summary scores: Physical Health Summary Score and Psychosocial Health Summary Score.
Change From Baseline in the Pediatric Migraine Disability Assessment (PedMIDAS) Total Score | Baseline (Week 0) through Week 12
  The PedMIDAS scale evaluates the impact of headache on school performance, disability at home and social/sport function. The score is a composite of the total of 6 questions.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (58):
- United States (31):
  - Rehabilitation & Neurological Services /ID# 270782, Huntsville, Alabama
  - Preferred Research Partner, Inc /ID# 270389, Little Rock, Arkansas
  - Preferred Research Partners /ID# 270419, Little Rock, Arkansas
  - Advanced Research Center /ID# 270257, Anaheim, California
  - Neuro Pain Research Center /ID# 271048, Fresno, California
  - Accellacare - Long Beach /ID# 270398, Long Beach, California
  - Excell Research /ID# 270258, Oceanside, California
  - Lumos Clinical Research Center /ID# 270582, San Jose, California
  - Sunwise Clinical Research /ID# 270431, Walnut Creek, California
  - Northwest Florida Clinical Research Group, LLC /ID# 270833, Gulf Breeze, Florida
  - Auzmer Research /ID# 271158, Lakeland, Florida
  - My Preferred Research /ID# 270312, Miami, Florida
  - Encore Medical Research - Weston /ID# 271139, Weston, Florida
  - Pediatric Neurology & Epilepsy Center Of Central Florida - Winter Park /ID# 275263, Winter Park, Florida
  - Deaconess Midtown Hospital /ID# 270572, Evansville, Indiana
  - Michigan Headache & Neurological Institute /ID# 270942, Ann Arbor, Michigan
  - Proven Endpoints LLC /ID# 270269, Ridgeland, Mississippi
  - Cct Research - Papillion Research Center /ID# 270393, Papillion, Nebraska
  - Healthy Perspectives - Innovate Mental Health Services /ID# 270847, Nashua, New Hampshire
  - Dent Neurologic Institute - Amherst /ID# 270260, Amherst, New York
  - Headache Wellness Center /ID# 270568, Greensboro, North Carolina
  - Frontier Clinical Research - Scottdale /ID# 270854, Scottdale, Pennsylvania
  - Frontier Clinical Research - Smithfield /ID# 270849, Smithfield, Pennsylvania
  - Access Clinical Trials Inc /ID# 270280, Nashville, Tennessee
  - UT Health Austin at Dell Childrens Neurology Clinic /ID# 270577, Austin, Texas
  - Earle Research /ID# 270424, Houston, Texas
  - Clinpoint Trials /ID# 270261, Waxahachie, Texas
  - Pantheon Clinical Research /ID# 270259, Bountiful, Utah
  - Alpine Research Organization - Clinton /ID# 276527, Clinton, Utah
  - Highland Clinical Research /ID# 270281, Salt Lake City, Utah
  - Frontier Clinical Research - Kingwood /ID# 271053, Kingwood, West Virginia
- Canada (2):
  - London Health Sciences Centre - Victoria Hospital & Children's Hospital /ID# 270659, London, Ontario
  - McGill University Health Centre - Glen Site. /ID# 270662, Montreal, Quebec
- Denmark (2):
  - Herlev Hospital /ID# 270482, Herlev, Capital Region
  - Regionshospitalet Godstrup /ID# 270481, Herning, Central Jutland
- Hungary (2):
  - Semmelweis Egyetem /ID# 271219, Budapest
  - Rozsavolgyi Rendelo-Ceba Bt. /ID# 271500, Budapest
- Italy (2):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 270756, Milan, Milano
  - Ospedale Pediatrico Bambino Gesù /ID# 270759, Rome, Roma
- Japan (8):
  - Konan Medical Center /ID# 270486, Kobe, Hyōgo
  - Umenotsuji Clinic /ID# 270484, Kochi, Kochi
  - Tominaga Clinic - Osaka /ID# 270483, Osaka, Osaka
  - Tokyo Headache Clinic /ID# 271610, Shibuya-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 270487, Shinjuku-ku, Tokyo
  - Tendo Brain Clinic /ID# 271410, Tendo-shi, Yamagata
  - Nagaseki Headache Clinic /ID# 271699, Kai, Yamanashi
  - Tanaka Neurosurgery & Headache Clinic /ID# 271346, Kagoshima
- Netherlands (2):
  - Canisius-Wilhelmina Ziekenhuis /ID# 270374, Nijmegen, Gelderland
  - HagaZiekenhuis /ID# 270379, The Hague, South Holland
- Poland (5):
  - Clinical Research Center Medic-R /ID# 270235, Poznan, Greater Poland Voivodeship
  - Athleticomed Sp. z o.o /ID# 270243, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o /ID# 270238, Krakow, Lesser Poland Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny /ID# 270239, Wroclaw, Lower Silesian Voivodeship
  - OHA-MED sp. z o.o /ID# 270242, Warsaw, Masovian Voivodeship
- CMRC Headlands LLC /ID# 271300, San Juan, Puerto Rico
- United Kingdom (3):
  - Medway Maritime Hospital /ID# 271885, Gillingham, Kent
  - Royal Aberdeen Children's Hospital /ID# 271664, Aberdeen, Scotland
  - Stepping Hill Hospital-Stockport NHS foundation trust /ID# 271883, Stockport

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-712